CLINICAL TRIAL: NCT05961969
Title: A Feasibility Study of Robotic Transabdominal Top-down Intersphincteric Resection With Double-stapling Coloanal Anastomosis for Distal Rectal Cancer
Brief Title: Robotic Top-down Intersphincteric Resection
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202107066RINA
Record Dates: First submitted 2023-07-09; First posted 2023-07-27 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
Keywords: Intersphincteric resection (ISR); Transabdominal ISR; Top-down ISR; Transanal ISR; Rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing robotic Transabdominal Top-down Intersphincteric Resection: Patients undergoing robotic Transabdominal Top-down Intersphincteric Resection with Double-stapling Coloanal Anastomosis
  Interventions: Procedure: Robotic surgery

INTERVENTIONS:
Procedure: Robotic surgery — 1. Patients with rectal cancer.
  2. Patients will undergo robotic Transabdominal Top-down Intersphincteric Resection with Double-stapling Coloanal Anastomosis

SUMMARY:
The present study is to develop the novel robotic surgical technique and enhance the surgery quality for the treatment of distal rectal cancer.

DETAILED DESCRIPTION:
The intersphincteric resection (ISR) for the treatment of distal rectal cancer has been a complex two-step surgical procedure consisting of transabdominal mobilization of the anorectum and transanal bowel resection with handsewn coloanal anastomosis. The availability of robotic systems may facilitate the transabdominal approach, simplify the surgical procedures, and achieve better anorectal function for patients with distal rectal cancer requiring an ISR. Consecutive 40 patients with distal rectal cancer undergoing the single-step robotic transabdominal ISR with the intent-to-treat principle will be recruited. The risk factors for a failed transabdominal ISR were identified from the prospectively maintained clinicopathologic data using univariate and multivariate analysis. The surgical outcomes, the anorectal function, and the tumor recurrence were compared between patients with a successful or failed robotic transabdominal ISR. The investigators believe that the present project can facilitate the development of the novel robotic surgical technique and enhance the surgery quality for the treatment of distal rectal cancer in our hospital and even in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* cT1-3 or yT 1-3 rectal adenocarcinoma whose low border was located below the anorectal sling (4 cm from anal verge), in which the required surgery meets the definition of ISR;
* Clinically Tumor-Node-Metastasis (TNM) stage I-III rectal adenocarcinoma;
* Curative and elective surgery;
* American Society of Anesthesiology (ASA) class Ⅰ to Ⅲ patients;
* Age between 20 and 75 years.

Exclusion Criteria:

* cT4 adenocarcinoma, i.e., the rectal cancer invaded to external sphincter or adjacent pelvic organs;
* Evidence of distant metastasis;
* Primary tumor mass≧8 cm in diameter;
* Morbidly obese patients, i.e., body mass index (BMI) ≧ 40 kg/m2 ;
* Previous major surgery of low upper abdomen;
* The adenocarcinoma has invaded to lateral pelvic side wall requiring a lateral pelvic lymph node dissection. (7) Patients with poor anorectal function (Wexner incontinence Score≧ 10)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients diagnosed as rectal cancer and met with the above inclusion and exclusion criteria will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Completion of transabdominal ISR | About one week
  1. The total mobilization and transection of anorectum was performed in the transabdominal down sequence, followed by the double-stapling technique for the coloanal anastomosis;
  2. the proximal and distal stapled tissue doughnuts recovered from EEA device were intact;
  3. A variable length of muscular cuff of proximal internal anal sphincter was removed with a TME specimen;
  4. To define a successful transabdominal total ISR, besides the above-mentioned three criteria, the anastomotic site should be checked by immediate anoscopy to confirm the stapling line is approximately at the level of anal intersphincteric groove.

SECONDARY OUTCOMES:
Circumferential resection margin (CRM) | About one week
  The radicality of CRM will be evaluated by a pathologist for any tumor invasion
Distal and proximal resection margin | About one week
  The radicality of distal and proximal margin
Length of operation time | Through the completion of surgery, an average of 5 hours
  The duration between skin incision and wound dressing
Length of postoperative ileus | 30 days
  One of the most common postoperative complication
Hospitalization | After patients' discharge from hospital, an average of 7 days
  The total days of stay in hospital during postoperative period
Degree of postoperative pain | After patients' discharge from hospital, an average of 7 days
  The visual analogue scale
Intraoperative complications | Within 5 hours
  Any adverse effect will be recorded.
The wound infection | 30 days
  the presence of thin discharge or local abscess in the operative wound, followed by the confirmation with Gram stains or bacterial cultures.
Acute anastomotic leakage | 30 days
  The presence of clinical features of peritonitis and bowel contents in the drainage during hospitalization.
Chronic anastomotic leakage | 6 months
  a defect at the anastomotic site that results in a communication with the bowel lumen.
Questionnaire to assess disability | 6 months
  Standardized questionnaire was given to patients to assess disability that included the number of days until return to partial activity, full activity, and work on the basis of their subjective responses.
Fecal incontinence | 6 months
  Wexner score, also known as Cleveland Clinic Fecal Incontinence Severity Scoring System (CCIS) is a fecal incontinence score from 0-20; where 0 is perfect continence and 20 is complete incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung LIANG, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- Jin-Tung LIANG, Taipei, Taiwan